CLINICAL TRIAL: NCT06061523
Title: A Phase I, Open-label, Randomized Crossover Study to Evaluate the Relative Bioavailability and the Effect of Food for Sotorasib Tablets in Healthy Participants
Brief Title: A Clinical Trial to Evaluate Bioavailability and Effect of Food for Sotorasib in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: FDA and EMA agreed existing data are appropriate for approval and no further BE studies are required.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20220098
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Healthy Participants
Keywords: Sotorasib; AMG 510
MeSH Terms: interventions — sotorasib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence ABC (Experimental): Participants will be administered sotorasib orally in the following order:
  Treatment A - as 4 tablets under fasting conditions (test) Treatment B - as 8 tablets under fasting conditions (reference) Treatment C - as 4 tablets under fed conditions (test)
  Interventions: Drug: Sotorasib
- Treatment Sequence BAC (Experimental): Participants will be administered sotorasib orally in the following order:
  Treatment B - as 8 tablets under fasting conditions (reference) Treatment A - as 4 tablets under fasting conditions (test) Treatment C - as 4 tablets under fed conditions (test)
  Interventions: Drug: Sotorasib

INTERVENTIONS:
Drug: Sotorasib — Oral Tablet
  Other Names: AMG 510

SUMMARY:
The primary objectives of the study are to compare the pharmacokinetics (PK) and demonstrate relative bioavailability of sotorasib administered as 4 oral tablets (test) to sotorasib administered as 8 oral tablets (reference) and to assess the effect of food on the PK of sotorasib administered as 4 oral tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female participants, between 18 and 60 years of age (inclusive), at the time of Screening.
* Body mass index, between 18 and 32 kg/m2 (inclusive), at the time of Screening
* Females of nonchildbearing potential
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) as assessed by the Investigator (or designee).

Exclusion Criteria:

* Inability to swallow oral medication or history of malabsorption syndrome.
* History of hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee) and in consultation with the Sponsor.
* Poor peripheral venous access.
* History or evidence, at Screening or Check in, of clinically significant disorder, condition, or disease, including not otherwise excluded that, in the opinion of the Investigator (or designee), would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
* History or evidence of clinically significant arrhythmia at Screening, including any clinically significant findings on the ECG taken at Check-in.
* History suggestive of esophageal (including esophageal spasm, esophagitis), gastric, or duodenal ulceration or bowel disease (including but not limited to peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease, or irritable bowel syndrome), or a history of gastrointestinal surgery other than uncomplicated appendectomy and hernia repair. History of cholecystectomy is not permitted.
* Estimated glomerular filtration rate (eGFR) less than 70 mL/min/1.73 m² as calculated by the Modification of Diet in Renal Disease (MDRD) equation, at Screening or Check-in.
* ALT or AST > ULN, at Screening or Check-in.
* Thyroid-stimulating hormone outside normal range.
* Positive hepatitis B or hepatitis C panel and/or positive human immunodeficiency virus test, at Screening. Participants whose results are compatible with prior immunity (vaccination or prior infection) may be included.
* Use of any over-the-counter or prescription medications within 30 days or 5 half-lives (whichever is longer) before enrollment. Acetaminophen (paracetamol) (up to 2 g per day) for analgesia will be allowed. Hormone-replacement therapy (e.g., estrogen) will be allowed.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-09-09 (Estimated); Study Completion 2024-09-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Sotorasib | Approximately 9 days
Area Under the Plasma Concentration-time Curve from Time Zero to the Last Quantifiable Concentration (AUClast) of Sotorasib | Approximately 9 days
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of Sotorasib | Approximately 9 days

SECONDARY OUTCOMES:
Number of Participants who Experience a Treatment-emergent Adverse Event (TEAE) | Approximately 9 days
Number of Participants who Experience a Serious Adverse Event (SAE) | Up to approximately 39 days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com